CLINICAL TRIAL: NCT02254954
Title: A Single-center, Open-label, Phase 1 Study of Macitentan, Radiotherapy and Temozolomide Concurrent Therapy Followed by Maintenance Therapy With Macitentan and Temozolomide in Subjects With Newly Diagnosed Glioblastoma
Brief Title: Clinical Study on Macitentan, RT and TMZ Concurrent Therapy Followed by Maintenance Macitentan and TMZ in Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision due to low recruitment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-118
Record Dates: First submitted 2014-09-23; First posted 2014-10-02 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Glioblastoma
Keywords: glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — macitentan; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan in combination with RT & TMZ (Experimental): Escalating doses of macitentan in combination with RT and TMZ, and maintenance TMZ.
  Interventions: Drug: Macitentan in combination with RT and TMZ

INTERVENTIONS:
Drug: Macitentan in combination with RT and TMZ — Escalating doses of macitentan in combination with RT and TMZ, and maintenance TMZ.
  Other Names: Temodar (temozolomide [TMZ]); macitentan; Radiotherapy

SUMMARY:
This is a prospective, single-center, open-label, 3+3 dose escalation Phase 1 safety study. Adults with newly diagnosed GBM or gliosarcoma will receive macitentan in addition to the standard of care treatment for GBM. The study consists of a screening period, a treatment period, and a 30-day safety follow up period. The treatment period includes 6 weeks of concurrent therapy (macitentan+RT+TMZ), 4 weeks of monotherapy (macitentan) and 12 cycles of maintenance therapy (macitentan+TMZ). The study will end when the last treated subject has completed study treatment and the 30-day safety follow-up period.

The planned duration of the study is approximately 34-38 months depending on the number of dose levels and cohorts of subjects enrolled. Subject participation in the study will be for approximately 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age
* Histologically proven supratentorial GBM or gliosarcoma
* Use of effective contraception by women of childbearing potental.
* Use of effective contraception by fertile males with a female partner of childbearing potential.
* Interval of at least 3 weeks after biopsy or open surgery and able to begin study treatment.
* Result from a post-operative contrast-enhanced brain MRI within 72 hours after surgery or biopsy.
* Adequate bone marrow function
* Karnofsky Performance Score of at least 70.

Exclusion Criteria:

* Prior treatment for glioblastoma or gliosarcoma.
* Evidence of leptomeningeal spread of glibolastoma or gliosarcoma.
* Tumor foci below the tentorium or beyond the cranial vault.
* Evidence of recent hemorrhage on post-operative contrast enhanced brain MRI (except hemosiderin, resolving hemorrhage changes related to surgery, presence of punctuate hemorrhage in tumor).
* Aspartate aminotransferase or alanine aminotransferase > 3 times the upper limit of normal.
* Supine systolic blood pressure < 100 mmHg or diastolic blood pressure < 50 mmHg.
* Medical history of orthostatic hypotension.
* International normalized ratio > 1.5 on anticoagulant therapy, active bleeding on low molecular weight heparin, or chronic condition with a high risk of bleeding.
* Severe renal impairment.
* Severe hepatic impairment.
* Severe, active co-morbidity: (e.g. cardiac disease; respiratory disease; chronic hepatitis; hemtological and bone marrow diseases; severe malabsoprtion; human immunodeficiency virus).
* No concurrent strong CYP3A4 inducers or inhibitors.
* No investigational drug within 4 weeks of starting study treatment.
* Any life-threatening condition that could affect protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicities observed during the first 10 weeks of study treatment (i.e., 6 weeks of concurrent therapy with macitentan, RT and TMZ and 4 weeks of monotherapy with macitentan). | Start of treatment to week 10

SECONDARY OUTCOMES:
Plasma concentrations of endothelin-1 | Baseline, Weeks 2, 6, and 10
Plasma concentrations of macitentan and its metabolite | Baseline, Weeks 2 and 6
Area under the plasma concentration-time curve (AUCτ) for macitentan during one dosing interval for subjects treated with doses of macitentan 150 mg or higher | Week 4
Peak plasma concentration (Cmax) of macitentan during one dosing interval for subjects treated with doses of macitentan 150 mg or higher | Week 4
Time to reach peak plasma concentration (Tmax) of macitentan during one dosing interval for subjects treated with doses of macitentan 150 mg or higher | Week 4
Number of adverse events (per Common Terminology Criteria for Adverse Events [CTCAE] criteria, version 4.03]) leading to premature discontinuation of study treatment | Starting from first dose of concurrent therapy (i.e., macitentan, TMZ, RT) until the end of treatment plus 30 days of follow-up
Number of subjects with marked laboratory abnormalities or abnormal electrocardiogram (ECG) findings | Starting from first dose of concurrent therapy (i.e., macitentan, TMZ, RT) until the end of treatment plus 30 days of follow-up
Change from baseline in pulse rate, systolic & diastolic blood pressure | Starting from first dose of concurrent therapy (i.e., macitentan, TMZ, RT) until the end of treatment plus 30 days follow-up
Exploratory efficacy endpoint of proportion of subjects with progression free survival (PFS) at 6 and 12 months | 6 and 12 months after the start of treatment
Number of adverse events (per CTCAE] criteria, version 4.03]) as a measure of safety and tolerability. | Starting from first dose of concurrent therapy (i.e., macitentan, TMZ, RT) until the end of treatment plus 30 days of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Investigational Site Web Address — http://www.mdanderson.org